CLINICAL TRIAL: NCT00526149
Title: Multicenter Parallel Phase II Trial of BI 2536 Administered as One Hour IV Infusion Every 3 Weeks in Defined Cohorts of Patients With Various Solid Tumors. A New Drug Screening Program of the EORTC Network of Core Institutions (NOCI)
Brief Title: BI 2536 in Treating Patients With Recurrent or Metastatic Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-90061; EORTC-90061; EUDRACT-2006-004529-27; EORTC-90061-BI 1216.18
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer; Endometrial Cancer; Head and Neck Cancer; Melanoma (Skin); Ovarian Cancer; Sarcoma
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent breast cancer; stage IV breast cancer; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III ovarian epithelial cancer; recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult leiomyosarcoma; uterine leiomyosarcoma; adult alveolar soft-part sarcoma; adult angiosarcoma; adult desmoplastic small round cell tumor; adult epithelioid sarcoma; adult fibrosarcoma; adult liposarcoma; adult malignant fibrous histiocytoma; adult malignant mesenchymoma; adult neurofibrosarcoma; adult rhabdomyosarcoma; adult synovial sarcoma; endometrial stromal sarcoma; ovarian carcinosarcoma; ovarian sarcoma; recurrent uterine sarcoma; stage IV uterine sarcoma; recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Breast Neoplasms; Endometrial Neoplasms; Head and Neck Neoplasms; Melanoma; Ovarian Neoplasms; Sarcoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Ovarian Epithelial; Leiomyosarcoma; Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Fibrosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Malignant mesenchymal tumor; Neurofibrosarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Sarcoma, Endometrial Stromal | interventions — BI 2536; Chromatography, High Pressure Liquid; Mass Spectrometry

INTERVENTIONS:
Drug: BI 2536
Other: high performance liquid chromatography
Other: mass spectrometry
Other: pharmacological study

SUMMARY:
RATIONALE: BI 2536 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects and how well BI 2536 works in treating patients with recurrent or metastatic solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate if BI 2536 demonstrates antitumor activity in the selected tumor types.
* Further document its safety profile in the treated patient population.
* Describe the plasma concentration time-course following administration of a single administration of BI 2536 in patients with different tumor types using an appropriate population pharmacokinetic model.

OUTLINE: This is a multicenter study.

Patients receive BI 2536 IV over 1 hour on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Blood is collected periodically during study. Plasma samples are analyzed for pharmacokinetic studies by HPLC and tandem mass spectrometry.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Tumor-specific criteria:

* Head and neck cancer:

  * Histologically or cytologically proven squamous cell carcinoma of the head and neck (excluding nasopharyngeal primaries)
  * Patients presenting with new non-irradiated lesions in pre-irradiated field as target lesions are eligible
  * Recurrent or metastatic disease, no longer suitable for local therapy
  * Prior use of chemotherapy/chemoradiotherapy/EGFR inhibitors for the treatment of the primary disease/nonmetastatic disease is allowed
  * No prior chemotherapy for recurrent or metastatic disease

    * Prior treatment with EGFR inhibitor for metastatic advanced disease is allowed
* Breast cancer

  * Histologically proven recurrent or metastatic adenocarcinoma of the breast that failed prior taxane and anthracycline therapy
  * Patient must have had a minimum of one line and a maximum of 2 lines of chemotherapy treatment given either as adjuvant treatment or for recurrence/metastatic disease
  * Patients who do not qualify for Her-2-based therapy allowed
  * Hormone receptor status not specified
* Ovarian cancer

  * Histologically proven ovarian epithelial cancer
  * Metastatic or inoperable locally advanced disease
  * Patients either progressing under or relapsing within 6 months of completion of any line of platinum and taxane-based therapeutic regimen for advanced disease
* Soft tissue sarcoma

  * Histologically proven advanced and/or metastatic malignant soft tissue sarcoma of high or intermediate grade and one of the following histologies defined by the WHO classification 2002:

    * Leiomyosarcoma, adipocytic sarcoma, synovial sarcoma, and others
    * Fibroblastic (adult fibrosarcoma, myxofibrosarcoma, sclerosing epithelioid fibrosarcoma)
    * So-called fibrohistiocytic (pleomorphic malignant fibrous histiocytoma [MFH], giant cell "MFH", inflammatory "MFH")
    * Malignant glomus tumors
    * Skeletal muscles (rhabdomyosarcoma, alveolar or pleomorphic) excluding embryonic rhabdomyosarcoma
    * Vascular (epithelioid hemangioendothelioma, angiosarcoma)
    * Uncertain differentiation (synovial, epithelioid, alveolar soft part, clear cell, desmoplastic small round cell, extra-renal rhabdoid, malignant mesenchymoma, perivascular epithelioid cell tumour [PEComa], intimal sarcoma) excluding chondrosarcoma, Ewing tumors/primitive neuroectodermal tumor (PNET)
    * Malignant peripheral nerve sheath tumors
    * Malignant solitary fibrous tumors
    * Undifferentiated soft tissue sarcomas not otherwise specified
    * Other types of sarcoma (not listed as not eligible), if approved by the Study Coordinator (written or e-mail approval needed prior to registration)
  * Excluded are any of the following:

    * Embryonic rhabdomyosarcoma
    * Chondrosarcoma
    * Osteosarcoma
    * Ewing tumors/primitive neuroectodermal tumors
    * Gastrointestinal stromal tumor
    * Dermatofibrosarcoma protuberans
    * Inflammatory myofibroblastic sarcoma
    * Neuroblastoma
    * Malignant mesothelioma
    * Mixed mesodermal tumors of the uterus
  * Patients must have received no more than one combination or two single agents of chemotherapy regimen for advanced disease and treatment must have included an anthracycline if not medically contraindicated
* Melanoma

  * Histologically proven metastatic malignant melanoma
  * Ocular melanomas are excluded
  * Patients must either not have received any prior chemotherapy for recurrent /metastatic disease or have received one line of chemotherapy pending LDH ≤ 2 times upper limit of normal (ULN)

    * One prior line of immunotherapy is allowed

General criteria:

* Measurable disease, defined as unidimensionally measurable based on RECIST with a target lesion of at least 20 mm or 10 mm measured by spiral CT scan
* Documented progressive disease proven by imaging prior to study entry (i.e., progression should be documented by 2 imaging scans performed within the past 6 months prior to registration showing progression according to RECIST)
* No clinical evidence of brain metastases

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-2
* ANC ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 9 mg/dL
* Serum creatinine ≤ to 175 μmol/L
* Bilirubin ≤ 1.5 times ULN
* AST/ALT ≤ 2.5 times ULN (5 times ULN with liver metastases)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Absence of any psychological, familial, sociological, or geographical factors that would potentially hamper compliance with the study protocol and follow-up schedule
* No other previous or active malignancy for at least 5 years with the exception of cone-biopsied carcinoma of the cervix and adequately treated basal or squamous cell skin carcinoma
* No concomitant intercurrent illnesses including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with trial requirement or that are considered relevant for the evaluation of the efficacy or safety of the trial drug

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since administration of any prior systemic treatment for the current malignancy including treatment with chemotherapy, radiotherapy, immunotherapy, hormonal therapy, and treatment with monoclonal antibodies, or small molecule tyrosine kinase inhibitors and others
* No persistence of toxicities from prior anticancer therapy deemed clinically relevant
* No treatment with any other investigational drug within the past four weeks or within less than four half-life times of the investigational drug before treatment with the trial drug (whatever is the longest period)
* No major surgery within 4 weeks prior to the first treatment with the trial drug
* Concurrent treatment with corticosteroids, including prednisone and bisphosphonates, is allowed as long as the treatment started before entry into the study and as long as the dose is stable for two weeks prior to enrollment in the present trial
* Palliative radiotherapy may be given during the study for bone pain or for other reasons not due to progressive disease (e.g., bronchial obstruction, ulcerating skin lesions)

  * The irradiated area should be limited and should not involve more than 10% of the bone marrow
  * The irradiated area cannot be used for tumor response assessment
* No other concurrent investigational drugs
* No concurrent anti-tumor therapies such as chemotherapy, hormone therapy, gene therapy, tyrosine kinase inhibitors, or therapy with monoclonal antibodies or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Confirmed objective response rate (complete and partial responses) as defined by RECIST

SECONDARY OUTCOMES:
Clinical benefit as assessed by RECIST
Duration of response
Overall progression-free survival
Overall survival
Safety as assessed by CTCAE version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoffski, MD, MPH, Study Chair — University Hospital, Gasthuisberg
Locations (1):
- U.Z. Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Result] Schoffski P, Blay JY, De Greve J, Brain E, Machiels JP, Soria JC, Sleijfer S, Wolter P, Ray-Coquard I, Fontaine C, Munzert G, Fritsch H, Hanft G, Aerts C, Rapion J, Allgeier A, Bogaerts J, Lacombe D. Multicentric parallel phase II trial of the polo-like kinase 1 inhibitor BI 2536 in patients with advanced head and neck cancer, breast cancer, ovarian cancer, soft tissue sarcoma and melanoma. The first protocol of the European Organization for Research and Treatment of Cancer (EORTC) Network Of Core Institutes (NOCI). Eur J Cancer. 2010 Aug;46(12):2206-15. doi: 10.1016/j.ejca.2010.03.039. Epub 2010 May 13. PMID 20471824